CLINICAL TRIAL: NCT00427310
Title: A Clinical Trial to Evaluate the Postoperative Portal Vein Infusion of 5-Fluorouracil and Heparin in Patients With Resectable Adenocarcinoma of the Colon
Brief Title: Liver Infusions of Fluorouracil in Treating Patients With Dukes' A, Dukes' B, or Dukes' C Colon Cancer Undergoing Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Northern California Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSABP C-02
Record Dates: First submitted 2007-01-18; First posted 2007-01-29 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Colorectal Cancer
Keywords: stage I colon cancer; stage II colon cancer; stage III colon cancer; adenocarcinoma of the colon
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Fluorouracil; Observation; Heparin

ARMS (2):
- Arm 1: Postoperative 5 FU + sodium heparin (Experimental): Continuous portal vein infusion with 5 FU 600 mg/m2 + 5000 units sodium heparin per day given for a total of 7 consecutive days.
  Interventions: Drug: fluorouracil; Drug: sodium heparin
- Arm 2: Postoperative observation (Active Comparator)
  Interventions: Other: Observation

INTERVENTIONS:
Drug: fluorouracil
  Other Names: 5 FU
  Arms: Arm 1: Postoperative 5 FU + sodium heparin
Other: Observation
  Arms: Arm 2: Postoperative observation
Drug: sodium heparin
  Arms: Arm 1: Postoperative 5 FU + sodium heparin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether giving fluorouracil into the liver is more effective than no further treatment for patients with colon cancer undergoing surgery.

PURPOSE: This randomized phase III trial is studying giving infusions of fluorouracil into the liver in treating patients with Dukes' A, Dukes' B, or Dukes' C colon cancer undergoing surgery.

DETAILED DESCRIPTION:
OBJECTIVES: Determine whether adjuvant therapy with portal hepatic perfusion of 5-fluorouracil and sodium heparin effectively prolongs the disease-free interval and increases survival in patients undergoing curative resection of adenocarcinoma of the colon.

OUTLINE: Randomized study. Patients are randomized preoperatively; those randomized to Arm 1 begin therapy intraoperatively or within 6 hours of colonic resection. Arm 1: 5-Fluorouracil plus sodium heparin. Those randomized to Arm 2 receive no adjuvant therapy. Arm 2: observation (no further treatment).

PROJECTED ACCRUAL: 1,334 patients will be entered over a 4-year period.

ELIGIBILITY:
Inclusion Criteria:

* more than one synchronous primary colon tumor
* white blood cell (WBC) > 4000/cu.mm. and platelet count greater than or equal to 100,000/cu.mm.
* evidence of adequate renal (serum creatinine less than or equal to 1.5 mg%) and hepatic function (bilirubin less than or equal to 1.5 mg%; serum glutamic oxaloacetic transaminase (SGOT) less than or equal to 60 I.U./ml)
* performance status of 0, 1 or 2
* Patients with intestinal obstruction are eligible. Preliminary or complementary colostomy does not preclude entry of a patient provided randomization is carried out prior to the planned curative resection.
* The distal margin of the tumor must be greater than or equal to 12 cm from the anal verge as endoscopically measured with the patient in the knee-chest position.
* Carcinoembryonic antigen (CEA) must be performed pre-operatively but results need not be known at the time of randomization.

Exclusion criteria:

* malignant colon tumors other than carcinoma, i.e., sarcoma, lymphoma, etc.
* patients whose tumors demonstrate free perforation
* previous or concomitant malignancy, regardless of site - except patients with squamous or basal cell carcinoma of the skin, and carcinoma in situ of the cervix which have been adequately treated
* patients who have received prior treatment other than preliminary or complementary colostomy (radiation, chemotherapy or surgery) for their current malignancy.
* patients having tumors within 12 cm of the anal verge
* performance status of 3 or 4
* patients having non-malignant systemic disease (cardiovascular, renal, hepatic, etc.) which would preclude their being subject to the chemotherapy treatment option
* patients who are pregnant at the time of randomization
* patients with psychiatric or addictive disorders which would preclude obtaining informed consent
* patients who have multiple primary tumors involving both the colon and the rectum which would preclude them from being classified as having only colon cancer or only rectal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1158 (Actual)
Dates: Start 1984-03; Primary Completion 1989-09 (Actual); Study Completion 2001-02 (Actual)

PRIMARY OUTCOMES:
Disease free interval | From randomization up to 4 years.
  Evidence of treatment failure (presence of tumor in local/regional or distant sites, confirmed by either biopsy or other acceptable evidence.
Survival | From randomization up to 4 years.

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc

REFERENCES:
- [Background] O'Connell MJ, Lavery I, Yothers G, Paik S, Clark-Langone KM, Lopatin M, Watson D, Baehner FL, Shak S, Baker J, Cowens JW, Wolmark N. Relationship between tumor gene expression and recurrence in four independent studies of patients with stage II/III colon cancer treated with surgery alone or surgery plus adjuvant fluorouracil plus leucovorin. J Clin Oncol. 2010 Sep 1;28(25):3937-44. doi: 10.1200/JCO.2010.28.9538. Epub 2010 Aug 2. PMID 20679606
- [Background] Wilkinson NW, Yothers G, Lopa S, Costantino JP, Petrelli NJ, Wolmark N. Long-term survival results of surgery alone versus surgery plus 5-fluorouracil and leucovorin for stage II and stage III colon cancer: pooled analysis of NSABP C-01 through C-05. A baseline from which to compare modern adjuvant trials. Ann Surg Oncol. 2010 Apr;17(4):959-66. doi: 10.1245/s10434-009-0881-y. PMID 20082144
- [Background] Wilkinson NW, Yothers G, Lopa SH, et al.: Long-term survival results of surgery alone compared with surgery plus 5-fluorouracil and leucovorin for stage II and stage III colon cancer: pooled analysis of NSABP adjuvant trials C-01 through C-05. [Abstract] American Society of Clinical Oncology 2009 Gastrointestinal Cancers Symposium, 15-17 January 2009, San Francisco, CA. A-442, 2009.
- [Background] Kim GP, Colangelo LH, Wieand HS, Paik S, Kirsch IR, Wolmark N, Allegra CJ; National Cancer Institute. Prognostic and predictive roles of high-degree microsatellite instability in colon cancer: a National Cancer Institute-National Surgical Adjuvant Breast and Bowel Project Collaborative Study. J Clin Oncol. 2007 Mar 1;25(7):767-72. doi: 10.1200/JCO.2006.05.8172. Epub 2007 Jan 16. PMID 17228023
- [Background] Allegra CJ, Paik S, Colangelo LH, Parr AL, Kirsch I, Kim G, Klein P, Johnston PG, Wolmark N, Wieand HS. Prognostic value of thymidylate synthase, Ki-67, and p53 in patients with Dukes' B and C colon cancer: a National Cancer Institute-National Surgical Adjuvant Breast and Bowel Project collaborative study. J Clin Oncol. 2003 Jan 15;21(2):241-50. doi: 10.1200/JCO.2003.05.044. PMID 12525515
- [Background] Wolmark N, Colangelo L, Wieand S. National Surgical Adjuvant Breast and Bowel Project trials in colon cancer. Semin Oncol. 2001 Feb;28(1 Suppl 1):9-13. doi: 10.1016/s0093-7754(01)90245-3. PMID 11273592
- [Background] Dignam JJ, Colangelo L, Tian W, Jones J, Smith R, Wickerham DL, Wolmark N. Outcomes among African-Americans and Caucasians in colon cancer adjuvant therapy trials: findings from the National Surgical Adjuvant Breast and Bowel Project. J Natl Cancer Inst. 1999 Nov 17;91(22):1933-40. doi: 10.1093/jnci/91.22.1933. PMID 10564677
- [Background] Mamounas E, Wieand S, Wolmark N, Bear HD, Atkins JN, Song K, Jones J, Rockette H. Comparative efficacy of adjuvant chemotherapy in patients with Dukes' B versus Dukes' C colon cancer: results from four National Surgical Adjuvant Breast and Bowel Project adjuvant studies (C-01, C-02, C-03, and C-04). J Clin Oncol. 1999 May;17(5):1349-55. doi: 10.1200/JCO.1999.17.5.1349. PMID 10334518
- [Result] Wolmark N, Rockette H, Petrelli N, et al.: Long-term results of the efficacy of perioperative portal vein infusion of 5-FU for treatment of colon cancer: NSABP C-02. [Abstract] Proceedings of the American Society of Clinical Oncology 13: A-561, 194, 1994.